CLINICAL TRIAL: NCT06430710
Title: Tooth Borne Versus Temporary Anchorage Devices Based Intrusion Systems for the Correction of Anterior Deep Overbite;Oral Hygiene, Pain and Treatment Effect
Brief Title: Tooth Borne Versus Temporary Anchorage Devices (TAD) Based Intrusion Systems for the Correction of Anterior Deep Overbite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2H
Record Dates: First submitted 2024-05-10; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Deep Overbite
Keywords: Anterior deep bite; Intrusive arch; Miniscrews
MeSH Terms: conditions — Overbite | interventions — Tooth Movement Techniques

STUDY DESIGN:
Intervention Model Description: Sixteen patients with anterior deep over bite participated in two groups each group contains eight patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mninscrew (Experimental): Miniscrews for incisor intrusion
  Interventions: Device: Intrusion
- Intrusive arch (Experimental): Continuous arch technique for incisor intrusion
  Interventions: Device: Intrusion

INTERVENTIONS:
Device: Intrusion — 2 different methods for incisor intrusion

SUMMARY:
Compare the tooth borne versus fixed orthodontic intrusive system (TADs) for the correction of anterior deep overbite

DETAILED DESCRIPTION:
this study determined which method was more compliant, efficacy and comfortable. It was performed to evaluate intrusion of upper incisors with applying tooth borne system as Connecticut Intrusion Arch (CIA) and temporary anchorage devices (TADs) [miniscrew] and evaluate the dental and skeletal cephalometric effects of these intrusion methods on individuals with deep bite caused by supraocclusion of upper incisors. It also evaluated oral hygiene and pain sensation in the two groups during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Class I or Class II malocclusion with minimal crowding.
2. 70% to 100% overbite.
3. High lip line with gingival display on smiling and super-eruption of maxillary incisors.
4. All patients had permanent dentition with average to vertical growth pattern and curve of Spee of 4mm or less.

Exclusion Criteria:

1. Having missing teeth on the anterior maxillary area.
2. Any history of trauma or root canal treatment.
3. Previous orthodontic treatment.
4. Low lip line duing social smile.
5. Having any hormonal disorder or syndromes.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Measure distance of insicors intrusion | 2 years
  measure in mm the distance of apical movement

SECONDARY OUTCOMES:
Pain intensity | 8 months
  By unit on Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt